CLINICAL TRIAL: NCT04612387
Title: Assessing the Effectiveness of a 12-week Online Wellness Intervention in Medical Students: a Pre-Post Single-arm Interventional Study
Brief Title: Online Wellness Intervention in Medical Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00098576
Record Dates: First submitted 2020-10-27; First posted 2020-11-03 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2020-10

CONDITIONS: Stress, Psychological; Mind Body Therapy; Wellbeing
MeSH Terms: conditions — Stress, Psychological | interventions — Mind-Body Therapies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mind-body Intervention arm (Experimental): Online yoga, meditation and nutrition tips.
  Interventions: Behavioral: Mind-body therapy

INTERVENTIONS:
Behavioral: Mind-body therapy — Online yoga, meditation and nutrition tips.

SUMMARY:
Medical students are at high risk of stress. This project will test how well a 12-week stress reduction program works to reduce stress, anxiety and depression and improve well-being. The program is delivered online and each week is made of an introduction video, 7-8 minutes of yoga, 5-7 minutes of meditation and nutrition tips. At the beginning and the end of the 12-week research study, we will be using surveys to ask students about their stress, anxiety, depression, sense of control over their own life, quality of life, and pain levels. After the program, the research team will conduct interviews with the medical student to allow them to share their other feedback about the program. The researchers will also send surveys to the medical students one month after the program ends to asses their continued satisfaction with and adherence to the program.

ELIGIBILITY:
Inclusion Criteria:

- Medical students in any year of medical school

Exclusion Criteria:

* Hospital Anxiety and Depression Scale (HADS) Depression score >10
* Active psychosis
* Post-traumatic stress disorder or frequent suicidal ideation
* Major medical co-morbidity
* Inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-10-25 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale | 12 weeks
  The degree to which situations in one's life are appraised as stressful will be assessed using the Perceived Stress Scale. The minimum score is 0, the maximum score is 40, and higher scores indicate a worse outcome.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | 12 weeks
  The Patient Health Questionnaire (PHQ-9) will be used to measure depression. The minimum score is 0, the maximum is 27, and higher scores indicate a worse outcome.
Psychological Wellbeing Scale | 12 weeks
  The Psychological Wellbeing Scale will be sued to measure well being. Higher scores mean higher levels of psychological well-being
Five Facet Mindfulness Questionnaire | 12 weeks
  Mindfulness will be assessed using the Five Facet Mindfulness Questionnaire.
Hospital Anxiety and Depression Scale (HADS) | 12 weeks
  Depression and anxiety will be measured on the Hospital Anxiety and Depression Scale. The minimum value is 0, the maximum is 21, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada